CLINICAL TRIAL: NCT05967403
Title: Anaesthesia Depth Consistency and System Performance of a Hermetic Closed-loop Anaesthesia Delivery System: A Randomized Controlled Study
Brief Title: Performance Analysis of Hermetic Closed-loop Anesthesia Delivery System
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sir Ganga Ram Hospital (Other)
Responsible Party: Principal Investigator, Nitin Sethi, DNB, Senior Consultant, Institute of Anaesthesiology, Pain & Perioperative Medicine, Sir Ganga Ram Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: EC/05/23/2282
Record Dates: First submitted 2023-07-21; First posted 2023-08-01 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Anesthesia
Keywords: propofol; closed-loop; anesthesia
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Intervention Model Description: One hundred and fifty participants (75/group) aged 18-65 years, ASA physical status I-II, of either sex, and undergoing elective non-cardiac surgery of minimum 60-minutes duration recruitment will be randomly divided into one of the two groups:
  Group-1 [Conventional CLADS (CC) group, n= 75]: Anaesthesia will be induced and maintained with propofol administered using the automated conventional CLADS.
  Group-2 [Hermetic CLADS (HC) group, n= 75]: Anaesthesia will be induced and maintained with propofol administered using the hermetic CLADS.
Who Masked: Participant, Outcomes Assessor
Masking Description: Inside the operating, the attending anaesthesiologist will not be blinded to the technique utilized to administer general anaesthesia (GA) and the recovery parameters immediately after extubation. However, the postoperative patient recovery profile will be evaluated by an independent assessor blinded to the GA technique and peri-extubation profile.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional CLADS group (Active Comparator): Propofol administration rate will be controlled by a feedback loop facilitated by BIS monitoring using the conventional (prototype) closed-loop anaesthesia delivery system (CLADS). A BIS value of 50 will be used as the target point for induction and maintenance of anesthesia
  Interventions: Drug: Propofol
- Hermetic CLADS group (Active Comparator): Propofol administration rate will be controlled by a feedback loop facilitated by BIS monitoring using the hermetic closed-loop anaesthesia delivery system (CLADS).[(Clarity Medical Private Ltd., Mohali, Punjab India]. A BIS value of 50 will be used as the target point for induction and maintenance of anesthesia
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Propofol — Propofol administration rate will be controlled by a feedback loop facilitated by BIS monitoring using the conventional closed loop anaesthesia delivery system (CLADS). A BIS value of 50 will be used as the target point for induction and maintenance of anaesthesia.
  Arms: Conventional CLADS group
Drug: Propofol — Propofol administration rate will be controlled by a feedback loop facilitated by BIS monitoring using the hermetic closed loop anaesthesia delivery system (CLADS). A BIS value of 50 will be used as the target point for induction and maintenance of anaesthesia.
  Arms: Hermetic CLADS group

SUMMARY:
Total intravenous anaesthesia (TIVA) is now a preferred technique for providing general anaesthesia (GA) because of its various inherent advantages like reduced postoperative nausea and vomiting (PONV), improved quality of post-operative recovery, anti-inflammatory and antioxidant action, anti-neoplastic activity, analgesic action, and absence of greenhouse effect. The evolution and advancement in automated anaesthesia delivery systems particularly for propofol have made propofol-TIVA more efficient by removing the human interface for both rate and concentration adjustments. Automated computer-controlled closed loop anaesthesia device adjusts propofol delivery based on patient's frontal cortex electrical activity determined by bispectral index (BIS).

Closed loop anaesthesia delivery system (CLADS) is an indigenously developed patented (Patent no.502/DEL/2003 & US 9,108,013 B2) computer-controlled anaesthesia delivery system which works with feedback loop information elicited by BIS monitoring and delivers propofol TIVA to the patient via a non-TCI automated infusion pump. It has been an extensively used and validated in patients undergoing both cardiac and non-cardiac surgical procedures.

A new compact and upgraded version of CLADS is now available. This new version incorporates the anesthetic depth monitor, hemodynamic monitor, controller, user interface and actuator syringe pump into a single, compact and user-friendly module.

The investigators aim to conduct a prospective randomized pilot study comparing the new CLADS and older CLADS version with respect to: adequacy of anaesthesia depth maintenance, performance characteristic of propofol delivery system, propofol requirement, haemodynamics stability, recovery from anesthesia and postoperative sedation.

DETAILED DESCRIPTION:
Propofol total intravenous anaesthesia (TIVA) is a preferred technique for providing induction and maintenance of general anaesthesia (GA). As opposed to the conventional inhaled anesthetics for maintaining GA, propofol TIVA has several advantages, such as, lower incidence of postoperative nausea and vomiting (PONV), antinociceptive and anti-inflammatory action, anti-neoplastic activity, and most importantly, its environment disposition (no greenhouse effect); and therefore, has potential to replace inhaled vapors for GA.

The introduction of target-controlled infusion (TCI) pumps has allowed precision control in propofol delivery as compared to the conventional manually operated infusion pumps. In manually operated infusion pumps the clinician regulates the propofol infusion rate to achieve the desired anaesthesia depth, whereas TCI-pumps deliver propofol using inbuilt algorithms based on the pharmacokinetic (PK) and pharmacodynamic (PD) profile of propofol. Two of the most used PK-PD models for propofol delivery are the Marsh model and the Schneider model. Whereas in the Marsh model the user can set the desired target plasma concentration, Schneider model allows the user to set the desired target effect site concentration for achieving adequate depth of GA.

Over the last two decades the evolution and advancement in automated anaesthesia delivery systems, particularly for propofol administration, has made propofol-TIVA delivery more efficient by removing the human interface required for adjusting real-time propofol delivery, both rate and concentration of propofol. Automated anaesthesia delivery systems deliver propofol based on ascertaining frontal cortex electrical activity as determined by the processed electroencephalogram, the bispectral index (BIS) score. These devices regulate propofol delivery based on a feedback loop involving the BIS score (control variable) generated by the patient and the propofol infusion pump (actuator) and attempts to keep the values within a pre-assigned range, consistent with robust GA depth.

Closed loop anaesthesia delivery system (CLADS) is an indigenously developed patented (Patent no.502/DEL/2003 & US 9,108,013 B2) computer-controlled anaesthesia delivery system which works with feedback loop information elicited by BIS monitoring and delivers propofol TIVA to the patient via a non-TCI automated infusion pump. The basic control algorithm is based on the relationship between the infusion rates of propofol and BIS values, taking into consideration the pharmacokinetic variables, such as, drug distribution and clearance. The system updates the EEG data every 5-seconds and calculates the BIS error, a difference between the target BIS and the actual BIS value using the proportional-integral-derivative (PID) controller. During anaesthesia induction the target concentration is achieved in a stepwise manner with BIS feedback received every 5-seconds. During maintenance phase of anaesthesia, the propofol delivery is modified every 1-epoch of 30-seconds duration. In each epoch an average of initial 3-BIS values (of every 5-seconds) and average of last 3-BIS values (of every 5-seconds) are compared, and a trend assessment is made. If the trend indicates increasing BIS values, then higher propofol rate is delivered by the infusion pump (actuator) and vice-versa. The control algorithm is implemented using a personal computer (PC) with a Pentium 4 processor. The PC controls communication with the infusion pump (Pilot-C, Fresenius, Paris, France) and the vital sign monitor (AS5, Datex Ohmeda Division, GE Healthcare, Singapore) through RS 232 serial ports.

CLADS has been extensively used and validated for administering propofol TIVA in patients undergoing both cardiac and non-cardiac surgical procedures. In a multi-centric study on evaluation of anaesthesia delivery by CLADS, it was shown that CLADS maintains depth of anaesthesia with far more precision as compared to manual administration.

A new compact and upgraded version of CLADS (Clarity Medical Private Ltd., Mohali, Punjab Indiais now available. The new version integrates the anaesthetic depth as well as the hemodynamic monitor, the controller, the user interface and the actuator syringe pump into a single, compact and user-friendly module.

The investigators aim to conduct a prospective randomised pilot to compare the multiple connected-unit conventional CLADS with the hermetically unit-integrated CLADS version, with respect to, the adequacy of anaesthesia depth (primary objective); and, performance characteristic, propofol requirement, haemodynamic stability, recovery from anaesthesia and postoperative sedation of the delivery systems (secondary objectives).

ELIGIBILITY:
Inclusion Criteria:

* aged 18-65 years-
* ASA physical status I-II
* undergoing elective non-cardiac surgery of minimum 60-minutes duration

Exclusion Criteria:

* Uncompensated cardiovascular disease (e.g., uncontrolled hypertension, atrio- ventricular block, sinus bradycardia, congenital heart disease, reduced LV compliance, diastolic dysfunction).
* Hepato-renal insufficiency.
* Any history of neurological disorder (e.g., epilepsy) or brain trauma
* Uncontrolled endocrine diseases (e.g., diabetes mellitus, hypothyroidism).
* Known allergy/hypersensitivity to the study drug.
* History of any psychiatric disorder and/or drug dependence/substance abuse.
* Requirement of postoperative ventilation.
* Refusal to informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-12-09 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Anaesthesia depth consistency | From beginning of anaesthesia till 5- minutes post skin closure
  It will be determined by the percentage of the anaesthesia time during which the BIS remained +/- 10 of the target BIS of 50

SECONDARY OUTCOMES:
Performance characteristic of propofol delivery system | From beginning of anaesthesia till 5- minutes post skin closure
  It will be determined using the Varvel criteria parameter :median performance error (MDPE). This parameter is calculated by the computer software which analyses the intraoperative BIS data. This parameter have no unit of measurement. It's just an abstract number. Higher the value means worse performance of propofol delivery system. It is not a scale.
Performance characteristic of propofol delivery system | From start of anesthesia till 5- minutes post skin closure
  It will be determined using the Varvel criteria parameter: median absolute performance error (MDAPE).This parameter is calculated by the computer software which analyses the intraoperative BIS data. This parameter have no unit of measurement. Its just a abstract number.Higher the value means worse performance of propofol delivery system. It is not a scale.
Performance characteristic of propofol delivery system | From start of anesthesia till 5- minutes post skin closure
  It will be determined using the Varvel criteria parameter: wobble. This parameter is calculated by the computer software which analyses the intraoperative BIS data. This parameter have no unit of measurement. Its just a abstract number.Higher the value means worse performance of propofol delivery system. It is not a scale.
Performance characteristic of propofol delivery system | From start of anesthesia till 5- minutes post skin closure
  It will be determined using the Varvel criteria parameter: global score. It is calculated using the formula Median absolute performance error + wobble / percentage of the anesthesia time during which the BIS remained +/- 10 of the target BIS of 50. This parameter have no unit of measurement. Its just a abstract number.Higher the value means worse performance of propofol delivery system. It is not a scale.
. Propofol induction dose (mg/kg) | From start of propofol injection till 10-minutes intraoperatively
  Dose of propofol required for induction of anaesthesia
. Propofol maintenance dose (mg/kg/h) | From start of propofol injection till 5-minutes post skin closure
  Dose of propofol required for maintenance of anaesthesia
Time to loss of consciousness (measured in minutes) | From start of propofol injection till 10-minutes intraoperatively
  The time taken (in minutes) from starting propofol induction using CLADS till loss of verbal response.
Time to induction of anaesthesia (measured in minutes) | From start of propofol injection till 10-minutes intraoperatively
  The time taken (in minutes) from starting propofol induction using CLADS till a target BIS value of '50' is achieved
Intra-operative heart Rate (beats per minute) | From beginning of anaesthesia till 10 hours intraoperatively]
  Comparison of intra-operative heart rate between the study arms will be done
Intra-operative systolic , diastolic, and mean blood pressure (mmHg) | From beginning of anaesthesia till 10 hours intraoperatively]
  Comparison of intra-operative blood pressure- systolic, diastolic, and mean blood pressure between the study arms will be done
Early recovery from anaesthesia (measured in minutes) | From end of anaesthesia till 20-minutes postoperatively
  Time taken by the patient to open his/her eyes after discontinuation of anaesthesia will be noted
Early recovery from anaesthesia (measured in minutes) | From end of anaesthesia till 20-minutes postoperatively
  Time taken for tracheal extubation after discontinuation of anaesthesia will be noted
Postoperative sedation | From end of anaesthesia till 24-hours postoperatively
  Will be assessed using Modified Observer's assessment of alertness/sedation scale. The scale has a maximum value of '5', which refers to a fully awake patient and a minimum value of '0' which refers to a deeply sedated patient.

CONTACTS AND LOCATIONS:
Overall Officials: Nitin Sethi, DNB, Study Director — Sir Ganga Ram Hospital, New Delhi, INDIA; Amitabh Dutta, MD, PGDHR, Principal Investigator — Sir Ganga Ram Hospital, New Delhi, INDIA; Goverdhan D Puri, MD, PhD, Study Chair — Post Graduate Institute of Medical Education & Research, Chandigarh, India
Locations (1):
- Nitin Sethi, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No